CLINICAL TRIAL: NCT04760769
Title: 58-Week Open-label Trial of Tavapadon in Parkinson's Disease (TEMPO-4 Trial)
Brief Title: Open-label Trial in Parkinson's Disease (PD)
Acronym: TEMPO-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-PD-004; 2019-002952-17 (EudraCT Number)
Record Dates: First submitted 2021-02-12; First posted 2021-02-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
Keywords: Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tavapadon (Experimental): Participants will receive a Tavapadon tablet at a dose of 5 milligrams (mg) to 15 mg once daily (QD) orally during 58-week treatment period.
  Interventions: Drug: Tavapadon

INTERVENTIONS:
Drug: Tavapadon — Participants will receive Tavapadon at a dose of (5 to 15) mg QD, orally during a 58-week treatment period.
  Other Names: PF-06649751; CVL-751

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term administration of flexible doses of tavapadon in participants with Parkinson's Disease.

ELIGIBILITY:
Key Inclusion Criteria:

Rollover participants are eligible for the study if they met the following inclusion criteria:

* Participants who complete the 27-week double-blind Treatment Period of Trial CVL-751-PD-001 (NCT04201093) or Trial CVL-751 PD-003 (NCT04542499) or the 27-week double-blind Treatment Period and 10-day Safety/Withdrawal Assessment Period of Trial CVL-751-PD-002 (NCT04223193) and enter this trial within 72 hours after completing the last trial visit in the double-blind trial. Rollover participants from Trial CVL-751-PD-003 must continue to use levodopa/carbidopa (or levodopa/benserazide) for the duration of the trial.
* Sexually active men or women of childbearing potential must agree to use acceptable (at minimum) or highly effective birth control, or remain abstinent during the trial and for 4 weeks after the last dose of trial treatment.
* Participants who are capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.
* Participants who are willing and able to refrain from any PD medications that are not permitted by the protocol (including dopaminergic agents) throughout participation in the trial.
* Participant who, in the judgement of the investigator, demonstrated adequate compliance with the IMP and protocol requirements in the double-blind trial.

Key Exclusion criteria:

Rollover participants are excluded from the trial if any of the following met:

* Participants who do not enroll in this open-label trial within 72 hours after completing the last trial visit in the double-blind trial
* Participants who answer "yes" on the C-SSRS Suicidal Ideation Item 4 or Item 5 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan, or Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting the criteria for C-SSRS Item 4 or Item 5 occurred within the last 6 months, OR Participants who answer "yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting the criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Participants who, in the opinion of the investigator, present a serious risk of suicide.
* Participants who had previously been enrolled in this open-label trial and had subsequently withdrawn.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | 62 Weeks
  An AE is any untoward medical occurrence in a participant or clinical trial participant, temporally associated with the use of trial intervention, whether or not considered related to the trial intervention. Any AE occurring following the start of treatment or occurring before treatment but increasing in severity afterward were counted as treatment-emergent AE (TEAE). Clinically significant abnormalities in Clinical Laboratory Evaluations, Vital Signs, Physical and Neurological evaluations and ECGs will be reported as TEAEs.
Number of Participants Who Discontinued Study Treatment | 62 Weeks
  A participant may discontinue the study treatment due to any of the following reasons: adverse event, death, worsening of PD symptoms to such an extent that, in the judgement of the investigator, the participant requires additional anti-PD medications, treatment with a prohibited concomitant medication, noncompliance with the trial schedule or procedures, withdrawal of consent, pregnancy, investigator discretion.
Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale (QUIP-RS) | 58 Weeks
  QUIP-RS is a global screening instrument that assesses impulse control disorders (ICDs) and related disorders (punding, hobbyism, and dopamine dysregulation syndrome) in participants with PD. The QUIP-RS has 4 primary questions that pertain to commonly reported thoughts, urges/desires, and behaviors associated with ICDs, each of which is applied to 4 ICDs (compulsive gambling, buying, eating, sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). The QUIP-RS uses a 5-point Likert scale (score 0-4 [0 means "never" and 4 means "very often"] for each question) to gauge the frequency of behaviors. Scores for each ICD and related disorder range from 0 to 16, with a higher score indicating greater severity (frequency) of symptoms. The total QUIP-RS score for all ICDs and related disorders combined ranges from 0 to 112.
Epworth Sleepiness Scale (ESS) | 58 Weeks
  ESS is a scale that is intended to measure daytime sleepiness. It assesses the likelihood of dozing off or falling asleep in the following common situations: sitting and reading, sitting inactive in a public place as a passenger in a car for an hour or more without stopping for a break, lying down to rest when circumstances permit, sitting and talking to someone, sitting quietly after a meal without alcohol, and in a car while stopped for a few minutes in traffic or at a light. Each situation is rated as 0 = would never nod off, 1 = slight chance of nodding off, 2 = moderate chance of nodding off, or 3 = high chance of nodding off. A score greater than or equal to (> =) 10 indicates that the participant may need to get more sleep, improve sleep practices, or seek medical attention to determine why he or she is sleepy.
Columbia-Suicide Severity Rating Scale (C-SSRS) | 60 Weeks
  C-SSRS rates an individual's degree of suicidal ideation (SI) on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent." The scale identifies SI severity and intensity, which may be indicative of an individual's intent to commit suicide. C-SSRS SI severity subscale ranges from 0 (no SI) to 5 (active SI with plan and intent).
Study Medication Withdrawal Questionnaire (SMWQ) | 60 Weeks
  SMWQ is a questionnaire to assess withdrawal symptoms subsequent to completion of dosing with Investigational medicinal product (IMP). The SMWQ is a modification of the Amphetamine Withdrawal Questionnaire, in which the first question "Have you been craving amphetamine or methamphetamine?" is replaced with "Have you been craving the trial medication?" This change is intended to prevent bias by implying that the trial medication might be an amphetamine or amphetamine-like stimulant when presented with the survey. Participants will complete the SMWQ onsite when they are at a designated trial visit; on days when the participant is not onsite, they will complete the SMWQ remotely.
Change From Baseline in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts I, II and III | 60 Weeks
  The MDS-UPDRS is a multidimensional scale that assesses the motor and non-motor impacts of PD across 4 parts. Part I, non-motor aspects of experiences of daily living, comprises 13 items, 6 of which are rated by the physician (Part IA) and 7 of which are rated by the participant (Part IB). Part II, motor aspects of experiences of daily living, comprises 13 items that are rated by the participant. Part III, motor examination, comprises 18 items that are assessed by the investigator (resulting in 33 scores by location and lateralization). Part IV, motor complications, comprises 6 item (3 items for dyskinesia and 3 items for fluctuation) and requires the physician to use historical and objective information to assess dyskinesia and motor fluctuations. Each item of all the parts will be rated on a scale from 0 to 4 on which 0 = normal, 1=slight, 2=mild, 3=moderate, and 4=severe. Change from baseline in MDS-UPDRS parts I, II and III combined score will be assessed.
Change From Baseline in the Hauser diary | 58 Weeks
  The Hauser diary (Hauser et al, 2000) assesses participant-defined clinical status over a period of time and provides a tool for assessment of the change in "off" time and "on" time with troublesome dyskinesia (which is a more accurate reflection of clinical response than "off" time alone). The Hauser diary asks participants to rate their mobility for each 30-minute period and to record their status for the majority of the period in 1 of 5 categories as: "on" time without dyskinesia, "on" time with nontroublesome dyskinesia, "on" time with troublesome dyskinesia, "off" time, or asleep.
Change From Baseline in the EuroQol 5 Dimension 5 Level (EQ-5D-5L) Index | Baseline (Day 1), Weeks 32 and 58
  EQ-5D-5L is a survey instrument used for participant-reported outcome that measures health in 5 dimensions. The EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each has 5 levels of perceived problems (1 = no problem, 2 = slight problems, 3 = moderate problems, 4 = severe problems, 5 = extreme problems). Participant selects an answer for each of 5 dimensions considering the response that best matches his/her health "today". The digits for the 5 dimensions are combined into a 5-digit number that describes the participant's health state.
Change From Baseline in the EuroQol 5 Dimension 5 Level (EQ-5D-5L) Visual Analog Scores (VAS) | Baseline (Day 1), Weeks 32 and 58
  EQ-5D-5L VAS is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. The EQ-5D-5L VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE Inc., Study Director — AbbVie
Locations (130):
- United States (51):
  - Birmingham, Alabama, Birmingham, Alabama
  - Pheonix, Arizona, Phoenix, Arizona
  - Little Rock, Arkansas, Little Rock, Arkansas
  - Fountain Valley, California, Fountain Valley, California
  - Fresno, California, Fresno, California
  - Los Angeles, California, Los Angeles, California
  - Pasadena, California, Pasadena, California
  - Reseda, California, Reseda, California
  - Englewood, Colorado, Englewood, Colorado
  - Florida, United States, Adventura, Florida
  - Boca Raton, Florida, Boca Raton, Florida
  - Coral Springs, Florida, Coral Springs, Florida
  - Maitland, Florida, Maitland, Florida
  - Naples, Florida, Naples, Florida
  - Ocala, Florida, Ocala, Florida
  - Port Charlotte, Florida, Port Charlotte, Florida
  - Port Orange, Florida, Port Orange, Florida
  - Tampa, Florida, Tampa, Florida
  - Winter Park, Florida, Winter Park, Florida
  - Augusta, Georgia, Augusta, Georgia
  - Chicago, Illinois, Chicago, Illinois
  - Winfield, Illinois, Winfield, Illinois
  - Kansas City, Kansas City, Kansas
  - Lexington, Kentucky, Lexington, Kentucky
  - Scarborough, Maine, Scarborough, Maine
  - Boston, Massachusettes, Boston, Massachusetts
  - Lawrence, Massachusetts, Lawrence, Massachusetts
  - East Lansing, Michigan, East Lansing, Michigan
  - West Bloomfield, West Bloomfield, Michigan
  - Las Vegas, Nevada, Las Vegas, Nevada
  - Camden, New Jersey, Camden, New Jersey
  - Albany, New York, Albany, New York
  - Syracuse, New York, Syracuse, New York
  - Asheville, North Carolina, Asheville, North Carolina
  - Durham, North Carolina, Durham, North Carolina
  - Cincinnati, Ohio, Cincinnati, Ohio
  - Cleveland, Ohio, Cleveland, Ohio
  - Columbus, Ohio, Columbus, Ohio
  - Dayton, Ohio, Dayton, Ohio
  - Toledo, Ohio, Toledo, Ohio
  - Philadelphia, Pennsylvania, Philadelphia, Pennsylvania
  - Memphis, Tennessee, Memphis, Tennessee
  - Georgetown, Texas, Georgetown, Texas
  - Houston, Texas, Houston, Texas
  - Lubbock, Texas, Lubbock, Texas
  - Round Rock, Texas, Round Rock, Texas
  - Burlington, Vermont, Burlington, Vermont
  - Richmond, Virginia, Richmond, Virginia
  - Virginia Beach, Virginia, Virginia Beach, Virginia
  - Kirkland, Washington, Kirkland, Washington
  - Spokane, Washington, Spokane, Washington
- Australia (6):
  - Erina, New South Wales, Erina, New South Wales
  - Kogarah, Kogarah, New South Wales
  - Macquarie Park, New South Wales, Sydney, New South Wales
  - Woolloongabba, Queensland, Woolloongabba, Queensland
  - Clayton, Victoria, Clayton, Victoria
  - Parkville, Victoria, Parkville, Victoria
- Bulgaria (5):
  - Medical center VITA1, Pleven, Pleven
  - Pleven, Bulgaria, Pleven
  - Pleven, Pleven
  - Multiprofile Hospital, Sofia, Sofia
  - Sofia, Sofia
- Canada (2):
  - Ottawa, Ontario, Ottawa, Ontario
  - Toronto, Ontario, Toronto, Ontario
- Czechia (4):
  - Chocen, Choceň, Chocen
  - Prague, Czech Republic, Prague, Czech Republic
  - Prague,, Prague
  - Rychnov nad Kněžnou, Rychnov nad Kněžnou
- France (7):
  - Creteil,, Créteil, Creteil
  - Boulevard Pinel, Bron, Bron
  - Grenoble cedex, Grenoble
  - Nancy, Nancy
  - Nîmes cedex 09, Nîmes
  - Strasbourg, Strasbourg
  - Toulouse Cedex 9, Toulouse
- Germany (9):
  - Muenster, Münster, Muenster
  - Bad Homburg, Bad Homburg
  - Berlin, Berlin
  - Bochum, Bochum
  - Gera, Gera
  - Haag in Oberbayern, Haag in Oberbayern
  - Klinikum rechts der Isar der TU München, Munich
  - Muenchen, München
  - Stadtroda, Stadtroda
- Hungary (3):
  - Budapest, Budapest
  - Pecs, Pécs
  - Tatabanya, Tatabánya
- Israel (5):
  - Haifa, Haifa
  - Petah Tiqva, Petah Tikva
  - Ramat Gan, Ramat Gan
  - Shoham, Shoham
  - Tel Aviv, Tel Aviv
- Italy (8):
  - Ancona, Ancona
  - Cassino, Cassino
  - Milano, Italy, Milan
  - Milano, Milan
  - Padova, Padua
  - Pisa, Pisa
  - Rome, Rome
  - Torino, Torino
- Poland (10):
  - Cracow, Krakow, Cracow
  - Siemianowice Slaskie, Siemianowice Śląskie, Siemianowice Slaskie
  - Centrum Medyczne NEUROMED, Bydgoszcz
  - Katowice, Katowice
  - Kraków, Krakow
  - Krakow, Krakow
  - Lublin, Lublin
  - Centrum Medyczne Hope Clinic Sebastian Szklener, Lublin
  - Warsaw, Warsaw
  - Singua, Warsaw
- Serbia (4):
  - Belgrade, Serbia, Belgrade
  - Belgrade,, Belgrade
  - Belgrade, Belgrade
  - Belgrade, Kragujevac, Belgrade
- Spain (10):
  - Elche, Elche, Alicante
  - Barcelona, Barcelona
  - Sant Cugat del Vallés Barcelona, Barcelona
  - San Sebastian, Donostia / San Sebastian
  - Madrid, Madrid
  - Móstoles, Madrid, Madrid
  - Pamplona, Pamplona
  - Sevilla, Seville
  - Terrassa, Terrassa
  - Valencia, Valencia
- Ukraine (6):
  - Zaporiizhzhya, Zaporizhzhya, Zaporiizhzhya
  - Zaporozhya, Zaporizhzhya, Zaporozhya
  - Dnipro, Dnipro
  - Lviv, Lviv
  - Vinnitsa, Vinnitsa
  - Medical Center, Zaporizhzhya, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No